CLINICAL TRIAL: NCT05332704
Title: A Randomised, Multi-centre, Double-blind, Placebo-controlled, Single Ascending Dose, Multiple Dose Study to Assess Safety, Tolerability, PK, PD & Preliminary Efficacy of IV Doses of ONO-4685 in Patients With Plaque Psoriasis
Brief Title: Safety, Tolerability, PK, PD and Preliminary Efficacy of ONO-4685
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ONO-4685-02; 2021-002151-10 (EudraCT Number)
Record Dates: First submitted 2022-03-18; First posted 2022-04-18 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Plaque Psoriasis
Keywords: Psoriasis; ONO-4685; PD-1; Bi-specific antibody; PD-1 Receptor; PD-1 Agonist
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Intervention Model Description: This is a phase I, multi-centre study to assess the safety, tolerability, PK & PD of ONO-4685. This study consists of: Part A single ascending dose, Part B an assessment of multiple doses & Part C to undertake initial assessment of efficacy with multiple doses.
  The study will recruit patients, male & female, with mild or moderate psoriasis diagnosed for at least 6 months. Following screening activities, patients are admitted to a clinical unit 1 day ahead of dosing and will stay at the unit for 4 nights. For patients receiving multiple doses, they will attend the clinic on the day of dosing and will stay for 3 nights. All patients will be followed up, for up to 24 weeks from 1st dose.
  The study will recruit 6 patients per cohort for part A & B and 18 patients per cohort for part C. The overall active to placebo ratio will be 2:1.
Who Masked: Participant, Investigator
Masking Description: This is a double-blind study.
  The pharmacist will be unblinded and is responsible for preparing blinded drug for administration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Part A, Active (Experimental)
  Interventions: Drug: ONO-4685
- Part A, Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Part B, Active (Experimental)
  Interventions: Drug: ONO-4685
- Part B, Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Part C, Active (Experimental)
  Interventions: Drug: ONO-4685
- Part C, Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ONO-4685 — -Part A: Single ascending doses of ONO-4685 as a single IV dose (Cohort A1-A5).
  Arms: Part A, Active
Drug: Placebo — -Part A: Single ascending doses of placebo as a single IV dose (Cohort A1-A5).
  Arms: Part A, Placebo
Drug: ONO-4685 — -Part B: Multiple doses of ONO-4685 as IV doses over a 4-week treatment period (Cohort B1 and B2)
  Arms: Part B, Active
Drug: Placebo — -Part B: Multiple doses of placebo as IV doses over a 4-week treatment period (Cohort B1 and B2).
  Arms: Part B, Placebo
Drug: ONO-4685 — -Part C: Multiple doses of ONO-4685 as IV doses over a 4-week treatment period (Cohort C1 and C2).
  Arms: Part C, Active
Drug: Placebo — -Part C: Multiple doses of placebo as IV doses over a 4-week treatment period (Cohort C1 and C2).
  Arms: Part C, Placebo

SUMMARY:
This is an early phase study to assess the safety and tolerability of ONO-4685 in patients with psoriasis. In addition, the study will assess how the drug is distributed and eliminated by the body (pharmacokinetics) and how the drug affects the body (pharmacodynamics). This will be done by measuring the amount of drug in the blood and measuring other markers in the body that might have been affected by ONO-4685. The study will also look at preliminary information on whether ONO-4685 might be effective in treating psoriasis.

The study will be split into three parts. Part A will assess a single dose of ONO-4685 in small groups of patients, each group planned to receive a higher dose than the last group. In Part B and C, patients will receive multiple doses of ONO-4685 over a period of 4 weeks.

ELIGIBILITY:
Inclusion Criteria

* Subjects must be willing and able to participate in the study
* A diagnosis of plaque-type psoriasis for ≥6 months.
* Plaque-type psoriasis involving ≥3% of body surface area (BSA) (Parts B and C).
* Willing to provide skin biopsies (Parts B and C).
* Subjects in good health, as judged by medical history, medical examination, vital signs, ECG and clinical laboratory tests.
* Subjects willing to comply with the contraception and sperm and ova donation requirements of the protocol.

Exclusion Criteria

* Subjects with any clinically significant abnormality in screening tests.
* Guttate, erythrodermic or pustular psoriasis as sole or predominant form of the psoriasis, or other skin condition (eg eczema).
* Presence or history of alcohol or drugs abuse.
* Heavy smokers (more than 20 cigarettes or use more than ½ ounce (12.5 grams) of tobacco each day).
* Subjects have had any 'live' vaccines (excluding COVID-19 vaccine) during the 3 months before the first dose of study medicine.
* Subjects have had a first COVID-19 vaccine within 6 weeks or second and booster COVID-19 vaccinations within 2 weeks before the first dose of study medicine.
* Subjects have had any clinically significant disease or infection, including tuberculosis.
* Presence or history of malignancy (cancer) including lymphoproliferative disorders.
* Subject is pregnant, lactating, or breastfeeding.
* Subjects have received treatment with biologics in the last 3 months, immunosuppressant medicine or prescription medicine for psoriasis within 4 weeks before admission to the ward; have used phototherapy from 2 weeks before admission to the ward; have used highly potent or potent topical steroids within 2 weeks before admission to the ward.
* Subjects have used topical corticosteroids or Vitamin D analogues within 7 days before admission to the ward (Parts B and C).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-03-25 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2024-07-18 (Actual)

PRIMARY OUTCOMES:
Treatment emergent adverse events (TEAEs) by severity | End of Study (3 years)
  Number of participants with TEAEs. An adverse event is any untoward medical occurrence in a participant who receives study drug without regard to possible causal relationship.
Clinical laboratory tests | End of Study (3 years)
  Number of participants with clinical laboratory abnormalities (including haematology, clinical chemistry and urinalysis).
Cytokines | Up to day 8 post dosing day
  Number of participants with elevated cytokines.
Lymphocytes | End of Study (3 years)
  Number of participants with depleted lymphocytes.
Vital signs (blood pressure) | End of Study (3 years)
  Number of participants with clinically significant changes in vital signs (blood pressure)
Vital signs (respiration rate) | End of Study (3 years)
  Number of participants with clinically significant changes in vital signs (respiration rate)
Vital signs (temperature) | End of Study (3 years)
  Number of participants with clinically significant changes in vital signs (temperature)
Vital signs (pulse rate) | End of Study (3 years)
  Number of participants with clinically significant changes in vital signs (pulse rate)
ECG parameters | End of Study (3 years)
  Number of participants with ECG abnormalities.

SECONDARY OUTCOMES:
Pharmacokinetics (Ceoi) | Part A, Day 1 (day of dosing). Part B and C, Day 1 (day of first dose) and Day 15 or 22 (day of last dose) depending on weekly or bi-weekly dosing.
  Assessment of the observed plasma concentration of ONO-4685 at the end of infusion (eoi).
Pharmacokinetics, Cmax | Part A up to day 85, Part B and Part C up to day 113
  Assessment of the maximum observed plasma concentration of ONO-4685.
Pharmacokinetics, Tmax | Part A up to day 85, Part B and Part C up to day 113
  Assessment of the time of maximum plasma concentration of ONO-4685.
Pharmacokinetics, AUC last | Part A up to day 85
  Assessment of the area under the plasma ONO-4685 concentration-time curve from time 0 to time of the last quantifiable concentration.
Pharmacokinetics, AUCinf | Part A up to day 85
  Assessment of the area under the plasma ONO-4685 concentration-time curve from time 0 to infinity.
Pharmacokinetics, CL (Clearance) | Part A up to day 85
  Assessment of the plasma clearance of ONO-4685.
Pharmacokinetics, Vss | Part A up to day 85
  Assessment of the volume of distribution at steady state of ONO-4685
Pharmacokinetics, T1/2 | Part A up to day 85, and after the last dose administration (Day 15 or 22) in Part B and Part C up to day 113.
  Assessment of the terminal elimination half-life of ONO-4685 in plasma.
Pharmacokinetics, AUCtau | Part B and C, after first (Day 1) and last (Day 15 or 22) dose
  Assessment of the area under the plasma ONO-4685 concentration-time curve during the dosing interval.
Pharmacokinetics, Ctrough | Part B and C, prior to administration of each dose
  Assessment of the trough concentration of ONO-4685 in plasma.
Pharmacodynamics, lymphocytes | Part A up to day 85, Part B up to day 113, Part C up to day 169
  Assessment of total lymphocytes, including subsets CD4+ T cell, CD8+ T cell, B cell and NK cell.
Pharmacodynamics, immunoglobulin | Part A up to day 85, Part B up to day 113, Part C up to day 169
  Assessment of total immunoglobulin, IgA, IgG and IgM.
Pharmacodynamics, cytokines | Part A up to day 8, Part B and Part C up to day 8 post last dose
  Assessment of cytokines, including IL-2, IL-6, IL-10, TNF-α and INF-γ.
Immunogenicity, Anti-ONO-4685-antibodies (ADA) | Part A up to day 85, Part B and Part C up to day 113
  Assessment of antibodies generated to ONO-4685 to measure potential immunogenicity.
Efficacy, Psoriasis Area and Severity Index (PASI) | Part A up to day 85, Part B up to day 113, Part C up to day 169
  Assessment of change in PASI from baseline.
Efficacy, Psoriasis Area and Severity Index (PASI) 50 | Part A up to day 85, Part B up to day 113, Part C up to day 169
  Assessment of number of subjects that achieve PASI 50, a 50% reduction in PASI from baseline.
Efficacy, Psoriasis Area and Severity Index (PASI) 75 | Part A up to day 85, Part B up to day 113, Part C up to day 169
  Assessment of number of subjects that achieve PASI 75, a 75% reduction in PASI from baseline.
Efficacy, Psoriasis Area and Severity Index (PASI) 90 | Part A up to day 85, Part B up to day 113, Part C up to day 169
  Assessment of number of subjects that achieve PASI 90, a 90% reduction in PASI from baseline.
Efficacy, Target Plaque Severity Score (TPSS) | Part A up to day 85, Part B up to day 113, Part C up to day 169
  Assessment of change in TPSS from baseline.
Efficacy, Physician's Global Assessment (PGA) | Part A up to day 85, Part B up to day 113, Part C up to day 169
  Assessment of change in PGA from baseline.
Efficacy, Physician's Global Assessment (PGA) 0/1 | Part A up to day 85, Part B up to day 113, Part C up to day 169
  Assessment of the number of subjects that achieve PGA 0/1.
Efficacy, Physician's Global Assessment (PGA) 0/1 and a 2-point improvement | Part A up to day 85, Part B up to day 113, Part C up to day 169
  Assessment of the number of subjects that achieve PGA 0/1 and a 2-point improvement from baseline.
Efficacy, Body Surface Area (BSA) | Part A up to day 85, Part B up to day 113, Part C up to day 169
  Assessment of the change in plaque BSA from baseline
Patient Reported Outcome, Dermatology Life Quality Index (DLQI) | Part A up to day 85, Part B up to day 113, Part C up to day 169
  Assessment of the change in DLQI from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Study Director — Ono Pharmaceutical Co. Ltd
Locations (4):
- Arensia Exploratory Medicine Phase 1 Unit, Chisinau, Moldova
- Arensia Exploratory Medicine, Bucharest, Romania
- United Kingdom (2):
  - Hammersmith Medicines Research, London
  - Medicines Evaluation Unit, Manchester

IPD SHARING:
Plan to Share IPD: No